CLINICAL TRIAL: NCT00257673
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety and Efficacy of MEM 1003 in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Safety and Efficacy of MEM 1003 Versus Placebo in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memory Pharmaceuticals (Industry)
Responsible Party: Amy S. Domanowski, Ph.D., Head Regulatory Affairs, Memory Pharmaceuticals Corp.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEM 1003-004; NCT00605501 (obsolete NCT alias)
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Alzheimer's Disease
Keywords: Cognition; Alzheimer's; Cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Active 30 mg MEM 1003
  Interventions: Drug: MEM 1003
- B (Experimental): 90 mg MEM 1003
  Interventions: Drug: MEM 1003
- C (Placebo Comparator): Placebo for MEM 1003
  Interventions: Drug: Placebo for MEM 1003

INTERVENTIONS:
Drug: MEM 1003 — 30 mg twice a day
  Arms: A
Drug: MEM 1003 — 90 mg MEM 1003 twice a day
  Arms: B
Drug: Placebo for MEM 1003 — Placebo twice a day
  Arms: C

SUMMARY:
The purpose of this study is to determine in a 12-week treatment study if MEM 1003 is a safe and effective treatment for patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease is the leading cause of dementia and one of the most common diseases of the aging population. It is a chronic brain disease that involves gradual memory loss, decline in the ability to perform routine tasks, disorientation, difficulty in learning, loss of language skills, impairment of judgment, and personality changes in affected individuals. The neurodegenerative nature of the disease eventually leads to the failure of other organ systems and death.

Perturbations in calcium homeostasis in the central nervous system, such as those associated with Alzheimer's disease and aging as well as stroke and head trauma can result in an increase in intracellular levels of calcium (Ca2+). Increased levels of Ca2+ may lead to cellular dysregulation and cell death. The role of calcium in these neurodegenerative processes led to the hypothesis that controlling calcium levels may be beneficial, particularly where progressive neuronal damage results in cognitive dysfunction and memory loss.

MEM 1003 is the (+)-enantiomer of a dihydropyridine that has been optimized for central nervous system activity. It inhibits L-type Ca2+ channels and within the anticipated human dosing range has more benign cardiovascular effects than other DHP L-Type calcium channel modulators.

ELIGIBILITY:
Inclusion Criteria:

* standardized MMSE Score of 10 to 24 points
* diagnosis of probable Alzheimer's disease
* magnetic resonance imaging or computed tomography examination compatible with AD
* modified Hachinski Ischemia Score of less than or equal to 4
* currently receiving no AD therapy or currently receiving donepezil, rivastigmine, or galantamine

Exclusion criteria:

* head injury associated with cognitive impairment
* history of vascular dementia stroke, transient cerebral ischemic episodes, major depression, major psychotic disorder, or symptomatic postural hypotension
* treatment for Alzheimer's disease other than donepezil, rivastigmine, or galantamine; tacrine is not permitted in the last 30 days or memantine in the last 90 days
* treatment with calcium channel blockers or any investigational medications within the prior 30 days

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Change from baseline at wk 12

SECONDARY OUTCOMES:
Other Cognitive Assessments, activities of daily living, functional assessments and safety

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Murray, MD, PhD, Study Director — Memory Pharmaceutical Corp.
Locations (54):
- United States (54):
  - Northport, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Sun City, Arizona
  - El Centro, California
  - Riverside, California
  - San Francisco, California
  - Torrence, California
  - Hamden, Connecticut
  - Washington D.C., District of Columbia
  - Brooksville, Florida
  - Chiefland, Florida
  - Coral Springs, Florida
  - Deerfield Beach, Florida
  - Delray Beach, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Plantation, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Towson, Maryland
  - Fall River, Massachusetts
  - Saint Loius, Missouri
  - Berlin, New Jersey
  - Long Branch, New Jersey
  - Princeton, New Jersey
  - Ridgewood, New Jersey
  - Toms River, New Jersey
  - Albany, New York
  - Staten Island, New York
  - Morganton, North Carolina
  - Portland, Oregon
  - Colmar, Pennsylvania
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Spartanburg, South Carolina
  - Johnson City, Tennessee
  - Bedford, Texas
  - Bulverde, Texas
  - San Antonio, Texas
  - Midvale, Utah
  - Bennington, Vermont
  - Norfolk, Virginia
  - Spokane, Washington